CLINICAL TRIAL: NCT05552365
Title: Randomised Pilot Control Trial for Reducing Anxiety Problems Among Children Indicated to Have Developmental Language Disorder
Brief Title: Reducing Anxiety Problems Among Children Indicated to Have Developmental Language Disorder
Acronym: RAP-iDLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Shaun Goh Kok Yew, Lecturer, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RP 2/21 SG (2021-T1-001-011)
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Developmental Language Disorder and Language Impairment; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Language Development Disorders; Language Disorders; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical interview (ADIS) will be administered by assessors who will not be told which arm participants are. Participants will be told not to mention intervention arm status to assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): 8-session cognitive behavioural intervention adapted for children indicated to have developmental language disorder.
  Interventions: Behavioral: Adapted Cognitive Behavioural
- Treatment as Usual (Other): Participants are re-directed to mental health support services. All participants given a mental health brochure which has contact details of mental health services for children.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Adapted Cognitive Behavioural — 8-session cognitive behavioural intervention adapted for children indicated to have developmental language disorder. Intervention includes psychoeducative, bodily relaxation, graded exposure, cognitive restructuring and brainstorming. Adaptations include increasing the number of visual supports, use of physical objects to illustrate concepts in addition to language.
  Arms: Active Intervention
Other: Treatment as Usual — Participants given a mental health brochure with contact information, where they can access services provided by mental health support service providers.
  Arms: Treatment as Usual

SUMMARY:
This study aims to pilot a world-first intervention, a mental health intervention augmented for children indicated with developmental language disorder (DLD). It serves as a proof-of-concept of how existing observational studies on these topics at the Centre for Research in Child Development (c.f. Tran-Sen; Gibber) can be translated into interventions. Mental health problems here are defined as anxiety type problems of social anxiety, specific phobia, separation anxiety and generalised anxiety. DLD is defined as a marked difficulty in oral language in the absence of biomedical causes (Bishop et al., 2017). This randomised pilot answers three uncertainties in preparation for a future definitive randomised control trial (RCT).

DETAILED DESCRIPTION:
This pilot aims to answer three uncertainties for a future randomised control trial (RCT), namely (1) Is the proposed intervention's efficacy sufficient (2) Are the proposed methods of recruitment sufficient (3) Are the proposed measures of evaluation sufficient Hypotheses: (1) Piloted intervention is sufficient for definitive RCT as 90% confidence intervals contain expected improvement versus treatment-as-usual (2) Piloted recruitment methods are sufficient for definitive RCT as recruitment rate is >4/month, dropout rate<25%. (3) Piloted measures are sufficient for definitive RCT as rates of unusable data are <20% and reliability alpha >.70.

ELIGIBILITY:
Inclusion Criteria:

* Shows signs of elevated anxiety, fear or stress, as rated on anxiety measures conducted by this study
* Enrolled in Primary 1 to 6 in a Ministry of Education Primary School
* Signs of a language difficulty [Either one of the following]

  1. Existing clinical opinion/report of this when child >5 years old
  2. Score <10th percentile on language measures conducted by this study

Exclusion Criteria:

* Conditions which exclude Developmental Language Disorder (e.g. Autism, Intellectual Disability, Hearing Impairment, other biomedical conditions).
* Non-anxiety disorder as primary mental health disorder
* Currently receiving treatment for anxiety disorder (e.g. pharmacotherapy or psychotherapy).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS-IV; Brown et al., 2004) | Administered at post treatment which is a maximum of 4 weeks from final session
  The ADIS-IV is a semi-structured interview organised diagnostically to permit differential diagnoses of anxiety disorders. Its yields a severity rating (0 to 8) which is utilised here as the primary outcome

SECONDARY OUTCOMES:
Screen for child anxiety related emotional disorders (SCARED; Birmaher et al., 1999) | Administered at post treatment which is a maximum of 4 weeks from final session
  The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder. The child report scores (41 items) and parent report scores (41 items) of the SCARED will be utilised here.
Child Anxiety Life Interference Scale (CALIS; Lyneham, et. al., 2013) | Administered at post treatment which is a maximum of 4 weeks from final session
  CALIS is a 2-part scale that measures child's anxiety life interference from both the child's and parent's perspectives. The children scale is a 10-item self-reported questionnaire on questionnaire evaluating the interference to the child's life and to the parent's life. All the items are related to common daily activities. The items are rated on a 5-point Likert scale (0 = Not at all, 1 = Only a little, 2 = Sometimes, 3 = Quite a lot, 4 = A great deal), where the higher scores indicate high levels of interference. Scores from the child and parent version will be used here

OTHER OUTCOMES:
Child Outcome and Session Rating Scales (CORS; Duncan et al., 2003) | At the end of each of the 8-sessions (each session is expected to run for 60 - 90 mins) for the active intervention
  The CORS is targeted for children aged 6 to 12 and has the same format as the Outcome Rating Scales (Duncan et al.,2003). It is written in a child-friendly language, where the child uses the happy and sad faces to understand the scale (Duncan et al., 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Shaun KY Goh, PhD, Principal Investigator — NTU-NIE
Locations (1):
- Centre for Research in Child Development, OER, NIE-NTU, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project Description — https://nie.edu.sg/research/projects/project/rp-2-21-sg-(2021-t1-001-011)